CLINICAL TRIAL: NCT05996900
Title: Investigating the Neural Mechanisms of Repetitive Brain Stimulation With Invasive and Noninvasive Electrophysiology in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Iowa (Other); Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corey Keller, Principal Investigator, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11354-1; 1R01MH132074 (NIH)
Record Dates: First submitted 2023-07-18; First posted 2023-08-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Epilepsy
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- TBS via direct electrical stimulation (Active Comparator)
  Interventions: Device: Intracranial electrodes
- TBS via transcranial magnetic stimulation (Active Comparator)
  Interventions: Device: TMS
- Sham TBS via direct electrical stimulation (Sham Comparator)
  Interventions: Device: Intracranial electrodes
- Sham TBS via transcranial magnetic stimulation (Sham Comparator)
  Interventions: Device: TMS

INTERVENTIONS:
Device: Intracranial electrodes — Intracranial electrodes will be used for the delivery of invasive brain stimulation.
  Arms: Sham TBS via direct electrical stimulation; TBS via direct electrical stimulation
Device: TMS — TMS will be used for the delivery of noninvasive brain stimulation both before and after implantation electrode surgery.
  Arms: Sham TBS via transcranial magnetic stimulation; TBS via transcranial magnetic stimulation

SUMMARY:
Transcranial magnetic stimulation (TMS) is an effective treatment for depression, but clinical outcome is suboptimal, partially because investigators are missing biologically-grounded brain markers which show that TMS is modifying activity at the intended target in the brain. The goal of this proposal is to characterize the key markers of the brain's response to repeated doses of TMS with high resolution using invasive brain recordings in humans, and relate these brain markers to noninvasive recordings. These markers will improve the understanding of TMS and can be used to optimize and enhance clinical efficacy for depression and other psychiatric disorders.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an effective treatment for major depressive disorder, but remission rates are 20-40%, and ideal stimulation parameters are unknown. rTMS is thought to work by changing the synaptic strength of neurons. The ability of the brain to make these changes is referred to as plasticity. rTMS-induced changes are thought to build with successive treatment sessions, a process referred to as metaplasticity. While both plasticity and metaplasticity are well-established in single cell physiology, relevance to rTMS in humans remains unknown. To improve clinical efficacy, the investigators need to understand 1) the neural response to a single rTMS session (plasticity), 2) the neural response to repeated daily rTMS sessions (metaplasticity), and 3) whether computational models of plasticity based on single-cell physiology apply to human patients receiving rTMS for depression.

Goals of the study are to 1) establish a detailed mechanistic understanding of the brain changes during current rTMS treatment; 2) identify clinically meaningful electrophysiological biomarkers for rTMS treatment; 3) establish a computational model to help predict both brain and clinical changes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65
* Medication-refractory epilepsy requiring phase II monitoring
* Must have intellectual capacity to ensure adequate comprehension of the study and potential risks involved in order to provide informed consent
* No current or history of major neurological disorders other than epilepsy

Exclusion Criteria:

* Those with a contraindication for MRIs (e.g. implanted metal)
* Any unstable medical condition
* Neurological or uncontrolled medical disease
* Active substance abuse
* Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
TMS-iEEG change after one TBS session | 45 minutes
  Change in evoked response measured after a single TBS session for active and sham, by resting state iEEG (intracranial EEG) and/or sEEG (stereo EEG).

SECONDARY OUTCOMES:
ES-iEEG change after one TBS session | 45 minutes
  Change in evoked response measured after a single TBS session for active and sham, by resting state iEEG and/or sEEG.
ES-iEEG change between two sequential TBS sessions | 45 minutes
  Change in single-pulse evoked response, or cortico-cortical evoked potentials (CCEPs), measured between two sequential TBS sessions, by resting state iEEG and/or sEEG.
TMS-iEEG change between two sequential TBS sessions | 45 minutes
  Change in single-pulse evoked response, or cortico-cortical evoked potentials (CCEPs), measured between two sequential TBS sessions, by resting state iEEG and/or sEEG.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States